CLINICAL TRIAL: NCT05585164
Title: Engage & Connect: A Novel Social Reward Psychotherapy for Postpartum Depression
Brief Title: Engage & Connect: A Psychotherapy for Postpartum Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 22-04024696
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Engage & Connect (Experimental)
  Interventions: Behavioral: Engage & Connect (E&C)
- Symptom Review and Psychoeducation (Experimental)
  Interventions: Behavioral: Symptom Review and Psychoeducation (SRP)

INTERVENTIONS:
Behavioral: Engage & Connect (E&C) — Engage & Connect, is a remotely-delivered extension of Engage psychotherapy. It is aimed to increase engagement in rewarding social activities and in turn, reduce postpartum depression. In each session, the therapist will work with the patient to develop "action plans" to pursue rewarding social activities of their choice with the goal of reducing social isolation.
  Arms: Engage & Connect
Behavioral: Symptom Review and Psychoeducation (SRP) — SPR is a remotely-delivered intervention aimed to increase knowledge of postpartum depression and monitor mental health changes. In each session, the therapist will review the participant's symptoms and discuss information related to postpartum depression and changes after birth.
  Arms: Symptom Review and Psychoeducation

SUMMARY:
This randomized controlled trial compares a novel psychotherapy, Engage & Connect, with a Symptom Review and Psychoeducation intervention, tailored to reduce postpartum depression. The study includes 9-weeks interventions, delivered remotely. It will examine changes in social isolation, processing of social rewards and depression severity over 9 weeks of treatment.

DETAILED DESCRIPTION:
Postpartum depression is linked with decreased motivation to seek rewarding activities and enjoyment of pleasurable experiences. Social isolation and low perceived social support predict persistence of postpartum depression. Engagement in rewarding social activities with significant others may increase motivation and enjoyment, motivating utilization of a therapy that addresses social isolation and reward response. The investigators developed Engage & Connect (E&C), a 9-week psychotherapy program that focuses on increasing meaningful social activities with significant others. This study will be a pilot Randomized Controlled Trial that will compare the 9-week E&C course for mothers with postpartum depression with a Symptom Review and Psychoeducation condition (SRP) for mothers with postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

1. Up to 1 year post-delivery
2. Edinburgh Postnatal Depression Scale (EPDS) score ≥ 10.
3. Off antidepressants or on a stable dose of an antidepressant for 8 weeks and do not intend to change the dose in the next 10 weeks.
4. Capacity to provide consent for research assessment and treatment.
5. Speaks English proficiently

Exclusion Criteria:

1. Intent or plan to attempt suicide in the near future
2. Ongoing psychotherapy (no more than once every 8 weeks or during the duration of the intervention)
3. Active substance abuse or dependence
4. Severe fetal anomalies, stillbirth or infant death at time of enrollment for index pregnancy
5. History or presence of psychiatric diagnoses other than major depressive disorder without psychotic features, generalized anxiety disorder, persistent depressive disorder, or specific phobia.
6. Use of psychotropic drugs or cholinesterase inhibitors other than use of ≤ 0.5 mg of lorazepam daily up to seven times per week.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Change in Edinburgh Postnatal Depression Scale (EPDS) | the EPDS will be measured Weekly for 9 weeks
  Measure of depression Severity. Scores range from 0 (no depression severity) to 30 (high depression severity)

SECONDARY OUTCOMES:
Change in Behavioral Activation for Depression Scale (BADS) | Baseline, Early Treatment (Week 3), Mid-treatment (Week 6) and Post Treatment (Week 9)
  25-item measure self-report measure of behavioral activation. Scores range from 0 (very low behavioral activation) to 150 (high behavioral activation).
Change in Social Reward Processing on STAR task | Baseline, Early Treatment (Week 3), Mid-treatment (Week 6) and Post Treatment (Week 9)
  Performance on the "Social Task for Assessment of Reward" [STAR]. Measured by reaction time to social feedback during reward trials on the task. Higher values of reaction time indicate slower response to social feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Nili Solomonov, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No